CLINICAL TRIAL: NCT06282822
Title: Multimodal Ultrasound Radiomics Based on Shear Wave Elastography for Accurate Diagnosis of Heart Failure With Preserved Ejection Fraction: A Prospective Multicenter Study
Brief Title: Shear Wave Elastography for Diagnosis of Heart Failure With Preserved Ejection Fraction
Status: Not yet recruiting | Type: Observational
Sponsor: First Hospital of China Medical University (Other)
Responsible Party: Principal Investigator, Chunyan Ma, Professor, First Hospital of China Medical University
Other Study IDs: HFpEF-SWE
Record Dates: First submitted 2024-02-13; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Shear Wave Elastography; Heart Failure With Preserved Ejection Fraction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Transthoracic echocardiography — All enrolled patients underwent noninvasive transthoracic echocardiography.

SUMMARY:
The diagnosis of heart failure with preserved ejection fraction (HFpEF) is often complex. Echocardiography has the advantages of being a non-invasive, simple operation, low price, and high repeatability, and is of great value in the diagnosis of HFpEF. However, the current echocardiographic assessment of left ventricular diastolic dysfunction and elevated filling pressure is based on multi-parameter indirect judgment, and new parameters are urgently needed to achieve accurate judgment of left ventricular diastolic function and an accurate diagnosis of HFpEF. Myocardial stiffness refers to the ability of the myocardium to undergo stress and strain. It is an important part of the pathophysiology of cardiac diastolic dysfunction and an important parameter for clinical evaluation of the diastolic function of HFpEF. Shear-wave elastography is a novel ultrasound-based elastography technology. Based on the shear wave generated by the remote induction of the radiation force of the focused ultrasound beam, the hardness of myocardial tissue can be measured quantitatively, locally, and noninvasively, and the change in myocardial stiffness in patients with HFpEF can be directly reflected. Currently, no relevant studies have applied shear-wave elastography to the diagnosis of HFpEF. This study aims to identify changes in myocardial stiffness measured by shear-wave elastography in patients with HFpEF based on a multicenter study and apply myocardial stiffness parameters to the diagnosis of HFpEF.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old
2. Clear epidemiological and population characteristics of HFpEF
3. Symptoms and/or signs of heart failure
4. Echocardiographic examination of LVEF≥50%
5. Objective evidence of cardiac structural and/or functional abnormalities consistent with left ventricular diastolic dysfunction and/or elevated left ventricular filling pressure, including elevated levels of natriuretic peptides
6. HFpEF score ≥6 or HFA-PEFF score ≥5

Exclusion Criteria:

Any one item per patient was excluded from the study:

1. Arrhythmia.
2. ischemic heart disease.
3. Valvular heart disease or congenital heart disease with severe hemodynamic changes.
4. History of pacemaker implantation or other cardiac surgery.
5. Poor ultrasonic image quality cannot meet the parameter measurement and analysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with heart failure with preserved ejection fraction
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-10-31 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Shear wave velocity | Completed within 2 weeks of enrollment